CLINICAL TRIAL: NCT02775266
Title: Effect of Systemic Administration of ALA (Alpha Lipoic Acid) as an Adjunct to Scaling and Rootplaning on Serum Resistin Levels in Patients With Chronic Periodontitis and Type 2 Diabetes Mellitus
Brief Title: Effect of Antioxidant Intake on Resistin Levels In Patients With Gum Disease and Diabetes
Acronym: EARGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, kinnera surapaneni, PG student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00159
Record Dates: First submitted 2016-05-05; First posted 2016-05-17 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus; Periodontitis
MeSH Terms: conditions — Diabetes Mellitus; Periodontitis | interventions — Thioctic Acid; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALA + Scaling and Root planing (Active Comparator): Systemic antioxidant Alpha lipoic acid 1800mg/day in 3 divided doses for a period of 3 months(group B)
  Interventions: Other: Alpha lipoic acid; Procedure: Scaling and Root planing
- Scaling and root planing only (Placebo Comparator): Patients will receive scaling and root planning at baseline and 3 months(group A)
  Interventions: Procedure: Scaling and Root planing

INTERVENTIONS:
Other: Alpha lipoic acid — Scaling and root planing will be done at baseline and systemic antioxidant Alpha lipoic acid 1800mg/day in 3 divided doses for a period of 3 months.
  Arms: ALA + Scaling and Root planing
Procedure: Scaling and Root planing — Scaling and root planing will be done at baseline.

SUMMARY:
To evaluate the effectiveness of non surgical periodontal therapy in addition to antioxidant(ALA) on resistin levels in patients with type 2 diabetes and periodontal disease

DETAILED DESCRIPTION:
A total of 40 patients with diabetes and chronic periodontitis attending the department of periodontics will be recruited in the study. 40 subjects will be randomly divided into two groups(control group and test group with 20 subjects in each group). Clinical parameters such as gingival index, periodontal index, random blood sugar levels(RBS) and glycosylated hemoglobin levels (Hb1aC) will be recorded at baseline and after 3 months and 2ml of blood sample will be collected by venepuncture ( baseline and after 3 months) and stored in Ethylenediaminetetraacetic acid containing vials to identify the levels of resistin in the patients by Enzyme linked immunosorbent assay. Group A will receive Alpha lipoic acid at baseline for a period of 3 months. Both the groups will receive scaling and rootplaning at baseline.

ELIGIBILITY:
Inclusion Criteria: Diabetic patients with Chronic periodontitis.

-

Exclusion Criteria: Smokers, Pregnant & lactating women, Prior periodontal therapy within 3 months.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Serum Resistin Levels and HBAIC Levels | 3 months
  2ml of blood sample will be collected by venepuncture at baseline and after 3 months and will be assessed by ELISA stored in EDTA containing vials to identify the levels of resistin in the patients by ELISA.
  Glycosylated hemoglobin levels (Hb1aC) will be recorded at baseline and after 3 months and assessed by Spectrophotometer.

SECONDARY OUTCOMES:
Gingival Index | 3 months
  Gingival index was recorded with william's periodontal probe at baseline and after 3 months
Probing pocket depth | 3 months
  Were recorded with william's periodontal probe at baseline and after 3 months
Clinical Attachment levels | 3 Months
  Were recorded with william's periodontal probe at baseline and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kinnera Surapaneni, [MDS], Principal Investigator — PANINEEYA INSTITUTE OF DENTAL SCIENCES ROAD NO: 5, KAMALANAGAR DILSUKHNAGAR, HYDERABAD - 500060; Rekha R Koduganti, MDS Perio, Study Director — Professor&HOD Dept.of.Periodontics,PMVIDS
Locations (1):
- Mohans Diabetic Centre, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mealey BL, Oates TW; American Academy of Periodontology. Diabetes mellitus and periodontal diseases. J Periodontol. 2006 Aug;77(8):1289-303. doi: 10.1902/jop.2006.050459. PMID 16881798
- [Background] Pendyala G, Thomas B, Kumari S. The challenge of antioxidants to free radicals in periodontitis. J Indian Soc Periodontol. 2008 Sep;12(3):79-83. doi: 10.4103/0972-124X.44100. PMID 20142950